CLINICAL TRIAL: NCT05955092
Title: Exploring the Application of 3D Bioprinting Technology in Constructing Preclinical Models of Pancreatic Cancer for Drug Sensitivity Testing and Its Significance in Personalized Treatment
Brief Title: Exploring the Application of 3D Bioprinting for Personalized Treatment in Pancreatic Ductal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PDAC3DP001
Record Dates: First submitted 2023-07-04; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to test the application value of 3D bioprinting technology in personalized treatment of pancreatic cancer.

The main questions it aims to answer are:

* Can 3D bioprinting technology be successfully applied to establish preclinical models of pancreatic cancer?
* Can 3D bioprinted preclinical models of pancreatic cancer be applied to personalized treatment of pancreatic cancer?

Participants will have tumor tissue collected to extract primary tumor cells for the establishment of in vitro preclinical models, which will be used for drug sensitivity testing.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Diagnosed as colorectal cancer with or without liver metastases before
* Pathologically proven colorectal cancer after surgery

Exclusion Criteria:

* History of other malignancies or serious medical conditions
* Inability to provide independent informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with clinically and pathologically confirmed pancreatic ductal adenocarcinoma are considered potential candidates for this study. Clinical physicians will comprehensively document the medical history, including only patients above 18 years of age. Individuals with other malignant tumors or severe diseases will be excluded. Patients who are unable to provide independent informed consent will not be included in this study. All patients in this study will undergo adjuvant/neoadjuvant chemotherapy and surgical resection for the treatment of localized pancreatic ductal adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of Drug Sensitivity in In Vitro Tumor Models with Clinical Response in Patients | From enrollment to end within 2 weeks
  1. Evaluation of the efficacy of neoadjuvant therapy in clinical response using the internationally recognized Response Evaluation Criteria in Solid Tumors (RECIST) 1.1: Stable Disease (SD) and Partial Response (PR) are considered indicators of chemotherapy sensitivity (good response), while Progressive Disease (PD) is considered indicative of chemotherapy resistance (poor response).
  2. Drug sensitivity testing results were assessed using standardized IC50 values. The standardized IC50 values were treated as the testing variables, while the clinical response to chemotherapy was designated as the state variable. The ROC curves for both variables were analyzed, and the area under the curve (AUC) was calculated to assess their correlation. To analyze the correlation between the drug testing results and clinical prognosis, linear regression analysis was performed to evaluate the correlation between standardized IC50 values and patients' progression-free survival (PFS) values.

SECONDARY OUTCOMES:
Progression-free survival time (PFS) | Up to 2 years.
  The time from the start of postoperative adjuvant therapy to recurrence or death.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) can be accessed with reasonable requests via e-mail. IPD will be shared after the study is completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD data will available after the study is completed.
Access Criteria: Data can be accessed via e-mail with reasonable requests.

REFERENCES:
- [Background] Boj SF, Hwang CI, Baker LA, Chio II, Engle DD, Corbo V, Jager M, Ponz-Sarvise M, Tiriac H, Spector MS, Gracanin A, Oni T, Yu KH, van Boxtel R, Huch M, Rivera KD, Wilson JP, Feigin ME, Ohlund D, Handly-Santana A, Ardito-Abraham CM, Ludwig M, Elyada E, Alagesan B, Biffi G, Yordanov GN, Delcuze B, Creighton B, Wright K, Park Y, Morsink FH, Molenaar IQ, Borel Rinkes IH, Cuppen E, Hao Y, Jin Y, Nijman IJ, Iacobuzio-Donahue C, Leach SD, Pappin DJ, Hammell M, Klimstra DS, Basturk O, Hruban RH, Offerhaus GJ, Vries RG, Clevers H, Tuveson DA. Organoid models of human and mouse ductal pancreatic cancer. Cell. 2015 Jan 15;160(1-2):324-38. doi: 10.1016/j.cell.2014.12.021. Epub 2014 Dec 31. PMID 25557080
- [Background] Grossman JE, Muthuswamy L, Huang L, Akshinthala D, Perea S, Gonzalez RS, Tsai LL, Cohen J, Bockorny B, Bullock AJ, Schlechter B, Peters MLB, Conahan C, Narasimhan S, Lim C, Davis RB, Besaw R, Sawhney MS, Pleskow D, Berzin TM, Smith M, Kent TS, Callery M, Muthuswamy SK, Hidalgo M. Organoid Sensitivity Correlates with Therapeutic Response in Patients with Pancreatic Cancer. Clin Cancer Res. 2022 Feb 15;28(4):708-718. doi: 10.1158/1078-0432.CCR-20-4116. PMID 34789479
- [Background] Tiriac H, Belleau P, Engle DD, Plenker D, Deschenes A, Somerville TDD, Froeling FEM, Burkhart RA, Denroche RE, Jang GH, Miyabayashi K, Young CM, Patel H, Ma M, LaComb JF, Palmaira RLD, Javed AA, Huynh JC, Johnson M, Arora K, Robine N, Shah M, Sanghvi R, Goetz AB, Lowder CY, Martello L, Driehuis E, LeComte N, Askan G, Iacobuzio-Donahue CA, Clevers H, Wood LD, Hruban RH, Thompson E, Aguirre AJ, Wolpin BM, Sasson A, Kim J, Wu M, Bucobo JC, Allen P, Sejpal DV, Nealon W, Sullivan JD, Winter JM, Gimotty PA, Grem JL, DiMaio DJ, Buscaglia JM, Grandgenett PM, Brody JR, Hollingsworth MA, O'Kane GM, Notta F, Kim E, Crawford JM, Devoe C, Ocean A, Wolfgang CL, Yu KH, Li E, Vakoc CR, Hubert B, Fischer SE, Wilson JM, Moffitt R, Knox J, Krasnitz A, Gallinger S, Tuveson DA. Organoid Profiling Identifies Common Responders to Chemotherapy in Pancreatic Cancer. Cancer Discov. 2018 Sep;8(9):1112-1129. doi: 10.1158/2159-8290.CD-18-0349. Epub 2018 May 31. PMID 29853643
- [Result] Xie F, Sun L, Pang Y, Xu G, Jin B, Xu H, Lu X, Xu Y, Du S, Wang Y, Feng S, Sang X, Zhong S, Wang X, Sun W, Zhao H, Zhang H, Yang H, Huang P, Mao Y. Three-dimensional bio-printing of primary human hepatocellular carcinoma for personalized medicine. Biomaterials. 2021 Jan;265:120416. doi: 10.1016/j.biomaterials.2020.120416. Epub 2020 Sep 22. PMID 33007612
- [Result] Sun L, Yang H, Wang Y, Zhang X, Jin B, Xie F, Jin Y, Pang Y, Zhao H, Lu X, Sang X, Zhang H, Lin F, Sun W, Huang P, Mao Y. Application of a 3D Bioprinted Hepatocellular Carcinoma Cell Model in Antitumor Drug Research. Front Oncol. 2020 Jun 3;10:878. doi: 10.3389/fonc.2020.00878. eCollection 2020. PMID 32582546